CLINICAL TRIAL: NCT02751931
Title: An Open-label, Baseline-controlled, Multicenter, Phase 3 Dose-titration Study Followed by a Fixed-dose Observation Period to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Children and Adolescents From 3 to Less Than 18 Years of Age With Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)
Brief Title: Open-label Phase 3 Study With Mirabegron in Children From 3 to Less Than 18 Years of Age With Neurogenic Detrusor Overactivity
Acronym: Crocodile
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 178-CL-206A; 2015-002876-25 (EudraCT Number)
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Neurogenic Detrusor Overactivity
Keywords: Pediatrics; Urodynamics; Mirabegron; Phase 3; Neurogenic Detrusor Overactivity
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Children (3 to < 12 Years) (Experimental): Participants aged 3 to < 12 years received initial dose of 25 milligram (mg) of mirabegron orally once daily based on weight (pediatric equivalent dose of 25 mg (milligram) [PED25]) on day 1. At weeks 2, 4 or 8, participant's were up-titrated to the pediatric equivalent dose of 50 mg in adults [PED50], orally once daily based on the given dose titration criteria. Following week 24, participants stayed on their individual dose level until week 52 end-of-study (EOS) or end-of-treatment (EOT).
  Interventions: Drug: Mirabegron
- Adolescents (12 to < 18 Years) (Experimental): Participants aged 12 to < 18 years received initial dose of 25 mg of mirabegron orally once daily based on weight [PED25] on day 1. At weeks 2, 4 or 8, participant's were up-titrated to the pediatric equivalent dose of 50 mg in adults [PED50] orally once daily based on the given dose titration criteria. Following week 24, participants stayed on their individual dose level until week 52 EOS or EOT.
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Participants received initial dose of 25 mg of mirabegron PED25 orally once daily. At weeks 2, 4 or 8, participants were up-titrated to PED50 based on the given dose titration criteria. Following week 24, participants stayed on their individual dose level until week 52 EOS or EOT. Participants with a body weight >=35 kg received mirabegron tablets or body weight <35 kg received mirabegron oral suspension. At week 24, participants on mirabegron oral suspension could switch to tablets if the body weight became >=35 kg or participants on mirabegron tablets could switch to oral suspension if the body weight became <35 Kg or participants could switch to either of the dosage form for acceptability reasons after sponsor's prior approval and on a case-by-case basis. Mirabegron extended-release granules were reconstituted with water to prepare a mirabegron oral suspension of 8 mg/mL. Administration was via an oral syringe with a sip of water afterwards.
  Other Names: YM178; Myrbetriq; Betanis; Betmiga

SUMMARY:
The objective of the study was to evaluate the efficacy, safety, tolerability and pharmacokinetics of mirabegron after multiple-dose administration in the pediatric population.

DETAILED DESCRIPTION:
This was a phase 3, open-label, baseline-controlled, multicenter study. The study consisted of 3 periods: Pretreatment period: for a maximum of 28 days before baseline, including screening, washout (if applicable) and baseline.

Efficacy treatment period: beginning the day after baseline and continuing to week 24. Long-term safety period: beginning after week 24 and continuing to week 52 (end of study [EOS]), or to the end of treatment (EOT).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body weight of greater than or equal to 11 kg.
* Subject suffers from NDO confirmed by urodynamic investigation at baseline. The diagnosis of NDO must be confirmed by the presence of at least 1 involuntary detrusor contraction > 15 cm H2O from baseline detrusor pressure, and/or a decrease in compliance leading to an increase in baseline detrusor pressure of > 20 cm H2O.
* Subject has been using CIC for at least 4 weeks prior to visit 1/screening.
* Subject has a current indication for drug therapy to manage NDO.
* Subject is able to take the study drug in accordance with the protocol

Exclusion Criteria:

* Subject has a known genitourinary condition (other than NDO) that may cause overactive contractions or incontinence or kidney/bladder stones or another persistent urinary tract pathology that may cause symptoms.
* Subject has one of the following gastrointestinal problems: partial or complete obstruction, decreased motility such as paralytic ileus, subjects at risk of gastric retention.
* Subject has a urinary indwelling catheter within 4 weeks prior to visit 1/screening.
* Subject has a surgically treated underactive urethral sphincter
* Subject has vesico-ureteral reflux grade 3 to 5.
* Subject has undergone bladder augmentation surgery.
* Subject receives electrostimulation therapy, if started within 30 days before visit 1/screening or is expected to start during the study period. Subjects who are on an established regimen may remain on this for the duration of the study.
* Subject suffers from a symptomatic urinary tract infection (UTI) at baseline (symptomatic is defined as pain, fever, hematuria, new onset foul-smelling urine). If present at visit 1/screening or diagnosed between visit 1/screening and visit 3/baseline, the UTI should be treated successfully (clinical recovery) prior to baseline. If a symptomatic UTI is present at baseline, all baseline assessments are allowed to be postponed for a maximum of 7 days until the UTI is successfully treated (clinical recovery).
* Subject has a (mean) resting pulse rate > 99th percentile [Fleming et al, 2011].
* Subject has an established hypertension and a systolic or diastolic blood pressure greater than the 99th percentile of the normal range determined by sex, age and height, plus 5mmHg [NIH 2005].
* Subject has a risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS]; or family history of LQTS, exercise-induced syncope).
* Subject has severe renal impairment (eGFR according to Larsson equation < 30 mL/min).
* Subject's aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is greater than or equal to 2 times the upper limit of normal (ULN) or total bilirubin (TBL) greater than or equal to 1.5 times the ULN according to age and sex.
* Subject has a history or presence of any malignancy prior to visit 1/screening.
* Subject has known or suspected hypersensitivity to mirabegron, any of the excipients used in the current formulations or previous severe hypersensitivity to any drug.
* Subject has participated in another clinical trial (and/or has taken an investigational drug within 30 days (or 5 half-lives of the drug, or the limit set by national law, whichever is longer) prior to visit 1/screening.
* Subject uses any of the following prohibited medications (after start of washout):

  * Any medication, other than the study drug used, for the management of NDO;
  * Any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index or sensitive P-glycoprotein (P-gp) substrates
  * Any strong CYP3A4 inhibitors if the subject has a mild to moderate renal impairment (eGFR 30 - 89 mL/min).
* Subject has been administered intravesical botulinum toxin; except if given > 4 months prior to visit 1/screening and the subject experiences symptoms comparable to those existing prior to the botulinum toxin injections.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Europe B.V.
Locations (32):
- Site AU61002, Randwick, New South Wales, Australia
- Belgium (2):
  - Site BE32004, Edegem
  - Site BE32001, Ghent
- Croatia (2):
  - Site HR38501, Zagreb
  - Site HR38503, Zagreb
- Denmark (2):
  - Site DK45001, Aarhus N
  - Site DK45002, Copenhagen
- Site IL97202, Jerusalem, Israel
- Jordan (2):
  - Site JO96202, Amman
  - Site JO96201, Irbid
- Site LV37101, Riga, Latvia
- Lithuania (2):
  - Site LT37002, Kaunas
  - Site LT37001, Vilnius
- Malaysia (2):
  - Site MY60001, George Town
  - Site MY60002, Kuala Lumpur
- Site MX52002, Mexico City, Mexico
- Site NO47001, Bergen, Norway
- Site PH63001, Quezon City, Philippines
- Poland (3):
  - Site PL48003, Gdansk
  - Site PL48001, Gdansk
  - Site PL48002, Warsaw
- Romania (2):
  - Site RO40002, Bucharest
  - Site RO40001, Bucharest
- Serbia (2):
  - Site RS38102, Niš
  - Site RS38101, Novi Sad
- Site SK42101, Bratislava, Slovakia
- South Korea (2):
  - Site KR82001, Seoul
  - Site KR82002, Seoul
- Site TW88601, New Taipei City, Taiwan
- Turkey (Türkiye) (3):
  - Site TR90002, Ankara
  - Site TR90006, Bursa
  - Site TR90008, Mersin

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Baka-Ostrowska M, Bolong DT, Persu C, Tondel C, Steup A, Lademacher C, Martin N. Efficacy and safety of mirabegron in children and adolescents with neurogenic detrusor overactivity: An open-label, phase 3, dose-titration study. Neurourol Urodyn. 2021 Aug;40(6):1490-1499. doi: 10.1002/nau.24657. Epub 2021 May 31. PMID 34058027
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;178-CL-206A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric participants consisting of male and female children from 3 to <12 years of age and adolescents from 12 to <18 years of age, with a body weight of >=11 kilogram (kg), with Neurogenic detrusor overactivity (NDO) on clean intermittent catheterization (CIC) were enrolled in this study.
Pre-assignment Details: Eligible participants who met inclusion and none of the exclusion criteria were enrolled. Participants who received oral drug to manage their NDO completed a 2 week washout period. A total of 113 pediatric participants were screened, 22 of whom were screening failures.
Groups:
- Children (3 to < 12 Years): Participants aged 3 to < 12 years received initial dose of 25 milligram (mg) of mirabegron orally once daily based on weight (pediatric equivalent dose of 25 mg (milligram) [PED25]) on day 1. At weeks 2, 4 or 8, participant's were up-titrated to the pediatric equivalent dose of 50 mg in adults [PED50] based on the given dose titration criteria. Following week 24, participants stayed on their individual dose level until week 52 end-of-study (EOS) or end-of-treatment (EOT).
- Adolescents (12 to < 18 Years): Participants aged 12 to < 18 years received initial dose of 25 mg of mirabegron orally once daily based on weight [PED25] on day 1. At weeks 2, 4 or 8, participant's were up-titrated to the pediatric equivalent dose of 50 mg in adults [PED50] based on the given dose titration criteria. Following week 24, participants stayed on their individual dose level until week 52 EOS or EOT.
Period: Overall Study
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Started | 56 | 35
Treated | 55 | 31
Completed | 43 | 27
Not Completed | 13 | 8
Not completed — Adverse Event | 3 | 0
Not completed — Other: Miscelleneous | 10 | 8

BASELINE CHARACTERISTICS:
Population: All Allocated Set included all participants who had a non-missing registration date at visit 3 (baseline).
Groups:
- Children (3 to < 12 Years): Participants aged 3 to < 12 years received initial dose of 25 mg of mirabegron orally once daily based on weight [PED25] on day 1. At weeks 2, 4 or 8, participant's were up-titrated to the pediatric equivalent dose of 50 mg in adults [PED50] based on the given dose titration criteria. Following week 24, participants stayed on their individual dose level until week 52 EOS or EOT.
- Total: Total of all reporting groups
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years) | Total
Number analyzed (Participants) | 56 | 35 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.9 (2.5) | 13.9 (1.6) | 10.2 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 15 | 48
  Male | 23 | 20 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 55 | 33 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 13 | 8 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 41 | 25 | 66
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Maximum Cystometric Capacity [Mean (Standard Deviation); unit: milliliter (mL)] — MCC was defined as the maximum bladder capacity reached during filling cystometry before either leakage or pain/discomfort was observed. Population: The analysis population consisted of the FAS (full analysis set) which included all participants who took >= 1 dose of study drug and provided both valid (as by the central reviewer's assessment) nonmissing MCC measurements at baseline and at a postbaseline visit for the primary efficacy endpoint.
  milliliter (mL)
    number analyzed (Participants) | 43 | 25 | 68
    (all) | 158.64 (94.50) | 238.92 (99.14) | 188.16 (103.15)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maximum Cystometric Capacity (MCC) at Week 24
Description: Change from baseline in MCC was based on filling urodynamics (volume at the end of filling). During urodynamic assessments, the bladder was filled until voiding/leakage began, or until the participant experienced pain or discomfort, or because dangerous high detrusor pressure, or 135% of maximum catheterized volume for age had been reached. A valid urodynamic assessment was confirmed valid by the central reviewers. Missing MCC observations at week 24 were imputed using last observation carried forward (LOCF).
Time Frame: Baseline and week 24
Population: The analysis population consisted of the full analysis set (FAS) which included all participants who took ≥ 1 dose of study drug and provided both valid (as by the central reviewer's assessment) nonmissing MCC measurements at baseline and at a postbaseline visit for the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Children (3 to < 12 Years): Participants aged 3 to < 12 years received initial dose of 25 mg of mirabegron orally once daily based on weight [PED25] on day 1. At weeks 2, 4 or 8, participant's were up-titrated to the pediatric equivalent dose of 50 mg in adults (PED50) based on the given dose titration criteria. Following week 24, participants stayed on their individual dose level until week 52 EOS or EOT.
- Adolescents (12 to < 18 Years): Participants aged 12 to < 18 years received initial dose of 25 mg of mirabegron orally once daily based on weight [PED25] on day 1. At weeks 2, 4 or 8, participant's were up-titrated to the pediatric equivalent dose of 50 mg in adults (PED50) based on the given dose titration criteria. Following week 24, participants stayed on their individual dose level until week 52 EOS or EOT.
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 43 | 25
mL | 72.09 (87.09) | 113.21 (82.99)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 72.09, 95% CI 2-sided [45.28 to 98.89]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 113.21, 95% CI 2-sided [78.95 to 147.47]

2. Secondary Outcome: Change From Baseline in Bladder Compliance (ΔV/ΔP)
Description: Bladder compliance was an indication of the elasticity of the bladder wall and was calculated by dividing the change in volume by the change in detrusor pressure during the filling of the bladder. Change from baseline in bladder compliance (change in volume/change in pressure) was assessed by the independent central reviewers and reported as annotations on the urodynamic trace and in an external database. During urodynamic assessments, the bladder was filled until voiding/leakage began, or until the participant experienced pain or discomfort, or because dangerous high detrusor pressure, or 135% of maximum catheterized volume for age had been reached. A valid urodynamic assessment was confirmed valid by the central reviewers.
Time Frame: Baseline and weeks 4 and 24
Population: The analysis population consisted of the FAS. Here, Overall Number of participants analyzed signifies number of participants evaluable for this outcome measure and number analyzed signifies number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mL/cm H2O
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 39 | 22
mL/cm H2O
  Change at Week 4 | -4.09 (50.78) | 15.16 (22.69)
  Change at Week 24: number analyzed (Participants) | 33 | 21
  Change at Week 24 | 14.62 (42.09) | 13.59 (15.02)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p = 0.618, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -4.09, 95% CI 2-sided [-20.55 to 12.38]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.005, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 15.16, 95% CI 2-sided [5.10 to 25.22]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.055, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 14.62, 95% CI 2-sided [-0.31 to 29.54]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 13.59, 95% CI 2-sided [6.75 to 20.42]

3. Secondary Outcome: Change From Baseline in Maximum Cystometric Capacity at Week 4
Description: Change from baseline in MCC was based on filling urodynamics (volume at the end of filling). During urodynamic assessments, the bladder was filled until voiding/leakage began, or until the participant experienced pain or discomfort, or because dangerous high detrusor pressure, or 135% of maximum catheterized volume for age had been reached. A valid urodynamic assessment was confirmed valid by the central reviewers.
Time Frame: Baseline and week 4
Population: The analysis population consisted of the FAS. Here, Overall Number of participants analyzed signifies those who where evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 41 | 23
mL | 41.36 (71.64) | 80.78 (96.15)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change from Baseline at week 4 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 41.36, 95% CI 2-sided [18.75 to 63.97]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 80.78, 95% CI 2-sided [39.20 to 122.36]

4. Secondary Outcome: Change From Baseline in Number of Overactive Detrusor Contractions (> 15 cm H20) Until End of Filling
Description: Detrusor overactivity is the occurrence of involuntary detrusor contractions during filling cystometry. During urodynamic assessments, the bladder was filled until voiding/leakage began, or until the participant experienced pain or discomfort, or because dangerous high detrusor pressure, or 135% of maximum catheterized volume for age had been reached. A valid urodynamic assessment was confirmed valid by the central reviewers.
Time Frame: Baseline and weeks 4 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: overactive detrusor contractions
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 41 | 22
overactive detrusor contractions
  Change at Week 4 | 0.44 (5.82) | -0.64 (2.94)
  Change at Week 24: number analyzed (Participants) | 36 | 22
  Change at Week 24 | -1.86 (4.16) | -0.77 (3.87)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p = 0.632, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.44, 95% CI 2-sided [-1.40 to 2.28]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.321, t-test, 2 sided; Mean Difference (Net) = -0.64, 95% CI 2-sided [-1.94 to 0.67]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.011, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -1.86, 95% CI 2-sided [-3.27 to -0.45]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.359, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -0.77, 95% CI 2-sided [-2.49 to 0.94]

5. Secondary Outcome: Change From Baseline in Detrusor Pressure at End of Filling
Description: Detrusor pressure was defined as bladder pressure minus intra-abdominal pressure as assessed by urodynamics. Filling was stopped (end of filling) when the detrusor pressure exceeded 100 cm H2O or was considered dangerously high by the investigator or urodynamicist (for instance, a prolonged passive detrusor pressure > 40 cm H2O). During urodynamic assessments, the bladder was filled until voiding/leakage began, or until the participant experienced pain or discomfort, or because dangerous high detrusor pressure, or 135% of maximum catheterized volume for age had been reached. A valid urodynamic assessment was confirmed valid by the central reviewers.
Time Frame: Baseline and weeks 4 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 41 | 22
cm H2O
  Change at Week 4 | -12.38 (19.56) | -6.48 (30.70)
  Change at Week 24: number analyzed (Participants) | 36 | 22
  Change at Week 24 | -18.11 (19.97) | -13.19 (19.91)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -12.38, 95% CI 2-sided [-18.56 to -6.21]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.334, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -6.48, 95% CI 2-sided [-20.09 to 7.13]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -18.11, 95% CI 2-sided [-24.87 to -11.35]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.005, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -13.19, 95% CI [-22.02 to -4.36]

6. Secondary Outcome: Change From Baseline in Filling Bladder Volume Until First Overactive Detrusor Contraction (> 15 cm H20)
Description: Detrusor overactivity is the occurrence of involuntary detrusor contractions during filling cystometry. During urodynamic assessments, the bladder was filled until voiding/leakage began, or until the participant experienced pain or discomfort, or because dangerous high detrusor pressure, or 135% of maximum catheterized volume for age had been reached. A valid urodynamic assessment was confirmed valid by the central reviewers. If no detrusor contraction of > 15 cm H2O occurred, the bladder volume was imputed with maximum cystometric capacity.
Time Frame: Baseline and weeks 4 and 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 21 | 8
mL
  Change at Week 4 | 54.00 [13.00 to 105.30] | 41.15 [3.00 to 62.50]
  Change at Week 24: number analyzed (Participants) | 13 | 8
  Change at Week 24 | 68.00 [32.00 to 110.0] | 62.00 [4.00 to 95.15]
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p < 0.001, Wilcoxon signed-rank test — From a Wilcoxon signed-rank test, testing the null hypothesis that week 4 median is equal to baseline median
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.148, Wilcoxon signed-rank test — From a Wilcoxon signed-rank test, testing the null hypothesis that week 4 median is equal to baseline median
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.002, Wilcoxon signed-rank test — From a Wilcoxon signed-rank test, testing the null hypothesis that week 24 median is equal to baseline median
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.039, Wilcoxon signed-rank test — From a Wilcoxon signed-rank test, testing the null hypothesis that week 24 median is equal to baseline median

7. Secondary Outcome: Change From Baseline in Filling Bladder Volume Until First Overactive Detrusor Contraction (> 15 cm H20): Wilcoxon Signed-rank Test Updated Analysis
Description: Detrusor overactivity is the occurrence of involuntary detrusor contractions during filling cystometry. During urodynamic assessments, the bladder was filled until voiding/leakage began, or until the participant experienced pain or discomfort, or because dangerous high detrusor pressure, or 135% of maximum catheterized volume for age had been reached. A valid urodynamic assessment was confirmed valid by the central reviewers. If no detrusor contraction of > 15 cm H2O occurred, the bladder volume was imputed with maximum cystometric capacity. This updated analysis is presented as the original analysis of bladder volume until first detrusor contraction (> 15 cm H2O) did not impute missing bladder volume data with the maximum cystometric capacity (MCC) value at that visit according to the statistical analysis plan (SAP). This analysis was updated to impute missing values for volume at first contraction with respective MCC values.
Time Frame: Baseline and weeks 4 and 24
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 41 | 24
mL
  Change at Week 4: number analyzed (Participants) | 41 | 23
  Change at Week 4 | 48.00 [5.00 to 88.00] | 46.30 [-23.90 to 176.00]
  Change at Week 24: number analyzed (Participants) | 38 | 24
  Change at Week 24 | 76.00 [32.00 to 147.20] | 78.45 [26.00 to 176.50]
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p < 0.001, Wilcoxon signed-rank test — From a Wilcoxon signed-rank test, testing the null hypothesis that week 4 median is equal to baseline median
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.007, Wilcoxon signed-rank test — From a Wilcoxon signed-rank test, testing the null hypothesis that week 4 median is equal to baseline median
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p < 0.001, Wilcoxon signed-rank test — From a Wilcoxon signed-rank test, testing the null hypothesis that week 24 median is equal to baseline median
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p < 0.001, Wilcoxon signed-rank test — From a Wilcoxon signed-rank test, testing the null hypothesis that week 24 median is equal to baseline median

8. Secondary Outcome: Change From Baseline in Filling Bladder Volume Until First Overactive Detrusor Contraction (> 15 cm H20): Paired T-test
Description: as for outcome 6
Time Frame: Baseline and weeks 4 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 41 | 24
mL
  Change at Week 4: number analyzed (Participants) | 41 | 23
  Change at Week 4 | 56.09 (96.23) | 73.80 (117.21)
  Change at Week 24: number analyzed (Participants) | 38 | 24
  Change at Week 24 | 93.09 (88.14) | 121.33 (159.84)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline was equal to 0
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.006, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline was equal to 0
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline was equal to 0
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline was equal to 0

9. Secondary Outcome: Change From Baseline in Average Catheterized Volume Per Catheterization
Description: For each participant, the average catheterized volume per catheterization was calculated as the sum of all available/non-missing catheterized volumes recorded over 2 measuring days in the weekend diary, whether or not the 2 days were consecutive divided by the number of catheterizations with non-missing volumes. If volumes were recorded on 1 single day of the weekend diary, the average catheterized volume per catheterization was calculated using all available/non-missing catheterized volumes recorded that day. If no volumes were recorded on any day of the weekend diary, the average catheterized volume per catheterization was missing. A valid bladder diary day in the weekend diary was any e-diary day for which ≥1 catheterized volume >0 mL was recorded with complete date and time.
Time Frame: Baseline and weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 43 | 24
mL
  Change at Week 2 | 14.58 (43.98) | 35.99 (54.19)
  Change at Week 4: number analyzed (Participants) | 42 | 24
  Change at Week 4 | 30.08 (49.50) | 51.96 (64.71)
  Change at Week 8: number analyzed (Participants) | 43 | 22
  Change at Week 8 | 36.90 (46.05) | 45.10 (53.77)
  Change at Week 12 | 32.25 (45.51) | 43.94 (58.49)
  Change at Week 24: number analyzed (Participants) | 41 | 23
  Change at Week 24 | 41.63 (58.03) | 59.31 (82.22)
  Change at Week 36: number analyzed (Participants) | 40 | 24
  Change at Week 36 | 53.87 (91.74) | 52.14 (74.90)
  Change at Week 52: number analyzed (Participants) | 40 | 23
  Change at Week 52 | 42.84 (65.31) | 42.40 (69.25)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 2 - Children; Test type: Other; p = 0.035, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 14.58, 95% CI 2-sided [1.0 to 28.1]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 2 - Adolescents; Test type: Other; p = 0.003, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 35.99, 95% CI 2-sided [13.1 to 58.9]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 30.08, 95% CI 2-sided [14.7 to 45.5]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 51.96, 95% CI 2-sided [24.6 to 79.3]
Statistical Analysis 5: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 8 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 36.90, 95% CI 2-sided [22.7 to 51.1]
Statistical Analysis 6: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 8 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 45.10, 95% CI 2-sided [21.3 to 68.9]
Statistical Analysis 7: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 12 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 32.25, 95% CI 2-sided [18.2 to 46.3]
Statistical Analysis 8: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 12 - Adolescents; Test type: Other; p = 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 43.94, 95% CI 2-sided [19.2 to 68.6]
Statistical Analysis 9: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 41.63, 95% CI 2-sided [23.3 to 60.0]
Statistical Analysis 10: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.002, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 59.31, 95% CI 2-sided [23.8 to 94.9]
Statistical Analysis 11: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 36 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 53.87, 95% CI 2-sided [24.5 to 83.2]
Statistical Analysis 12: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 36 - Adolescents; Test type: Other; p = 0.002, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 52.14, 95% CI 2-sided [20.5 to 83.8]
Statistical Analysis 13: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 52 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 42.84, 95% CI 2-sided [22.0 to 63.7]
Statistical Analysis 14: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 52 - Adolescents; Test type: Other; p = 0.008, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 42.40, 95% CI 2-sided [12.5 to 72.3]

10. Secondary Outcome: Change From Baseline in Maximum Catheterized Volume
Description: For each participant, the maximum catheterized volume per day was calculated using all available/non-missing catheterized volumes recorded for the 2 measuring days in the weekend e-diary, whether or not these 2 days were consecutive. Maximum value was calculated separately for each measuring day and the mean of the two values was used. If volumes recorded on 1 single day of the weekend e-diary, the maximum catheterized volume per day was calculated using all available/non-zero catheterized volumes recorded that day. If no volumes were recorded on any day of the weekend e-diary, the maximum catheterized volume per day was missing. A valid bladder diary day in the weekend diary was any e-diary day for which >=1 catheterized volume >0 mL was recorded with complete date and time.
Time Frame: Baseline and weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 43 | 24
mL
  Change at Week 2 | 17.50 (73.58) | 42.38 (78.23)
  Change at Week 4: number analyzed (Participants) | 42 | 24
  Change at Week 4 | 46.69 (80.29) | 73.25 (103.98)
  Change at Week 8: number analyzed (Participants) | 43 | 22
  Change at Week 8 | 45.27 (75.22) | 42.86 (79.97)
  Change at Week 12 | 33.23 (68.31) | 47.29 (69.83)
  Change at Week 24: number analyzed (Participants) | 41 | 23
  Change at Week 24 | 49.88 (103.70) | 84.39 (121.98)
  Change at Week 36: number analyzed (Participants) | 40 | 24
  Change at Week 36 | 60.09 (121.66) | 54.78 (104.54)
  Change at Week 52: number analyzed (Participants) | 40 | 23
  Change at Week 52 | 53.51 (96.72) | 54.30 (104.74)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 2 - Children; Test type: Other; p = 0.126, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 17.50, 95% CI 2-sided [-5.1 to 40.1]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 2 - Adolescents; Test type: Other; p = 0.014, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 42.38, 95% CI 2-sided [9.3 to 75.4]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 46.69, 95% CI 2-sided [21.7 to 71.7]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.002, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 73.25, 95% CI 2-sided [29.3 to 117.2]
Statistical Analysis 5: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 8 - Children; Test type: Other — Pre-Specified; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 45.27, 95% CI 2-sided [22.1 to 68.4]
Statistical Analysis 6: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 8 - Adolescents; Test type: Other; p = 0.020, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 42.86, 95% CI 2-sided [7.4 to 78.3]
Statistical Analysis 7: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 12 - Children; Test type: Other; p = 0.003, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 33.23, 95% CI 2-sided [12.2 to 54.3]
Statistical Analysis 8: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 12 - Adolescents; Test type: Other; p = 0.003, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 47.29, 95% CI 2-sided [17.8 to 76.8]
Statistical Analysis 9: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.004, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 49.88, 95% CI 2-sided [17.1 to 82.6]
Statistical Analysis 10: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.003, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 84.39, 95% CI 2-sided [31.6 to 137.1]
Statistical Analysis 11: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 36 - Children; Test type: Other; p = 0.003, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 60.09, 95% CI 2-sided [21.2 to 99.0]
Statistical Analysis 12: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 36 - Adolescents; Test type: Other; p = 0.017, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 54.78, 95% CI 2-sided [10.6 to 98.9]
Statistical Analysis 13: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 52 - Children; Test type: Other; p = 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 53.51, 95% CI 2-sided [22.6 to 84.4]
Statistical Analysis 14: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 52 - Adolescents; Test type: Other; p = 0.021, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 54.30, 95% CI 2-sided [9.0 to 99.6]

11. Secondary Outcome: Change From Baseline in Maximum Catheterized Daytime Volume (MCDV)
Description: For each participant, the MCDV was calculated using all available/non-missing catheterized daytime volumes for the 2 measuring days in the weekend e-diary, whether or not the 2 days were consecutive. Maximum value was calculated separately for each measuring day and the mean of the 2 values was used. If volumes were recorded on 1 single day of the weekend e-diary, the MCDV was calculated using all available/non-zero catheterized daytime volumes recorded that day. If no volumes were recorded on any day of the weekend e-diary, the MCDV was missing. Daytime was defined as the time between wake-up time (minus 30 min) & time to sleep (plus 29 min) recorded in the e-diary. A valid bladder diary day in the weekend diary was any e-diary day for which >=1 catheterized volume >0 mL was recorded with complete date and time.
Time Frame: Baseline and weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 43 | 24
mL
  Change at Week 2 | 18.13 (73.38) | 35.58 (86.78)
  Change at Week 4: number analyzed (Participants) | 42 | 24
  Change at Week 4 | 37.71 (83.33) | 70.35 (113.98)
  Change at Week 8: number analyzed (Participants) | 43 | 22
  Change at Week 8 | 43.91 (74.44) | 38.11 (90.88)
  Change at Week 12 | 29.05 (67.86) | 43.04 (73.82)
  Change at Week 24: number analyzed (Participants) | 41 | 23
  Change at Week 24 | 44.20 (98.31) | 81.37 (117.77)
  Change at Week 36: number analyzed (Participants) | 40 | 24
  Change at Week 36 | 58.49 (121.12) | 50.90 (114.05)
  Change at Week 52: number analyzed (Participants) | 40 | 23
  Change at Week 52 | 53.76 (100.24) | 49.13 (117.23)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 2 - Children; Test type: Other; p = 0.113, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 18.13, 95% CI 2-sided [-4.5 to 40.7]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 2 - Adolescents; Test type: Other; p = 0.056, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 35.58, 95% CI 2-sided [-1.1 to 72.2]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p = 0.005, t-test, 2 sided; From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 37.71, 95% CI 2-sided [11.7 to 63.7]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.006, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 70.35, 95% CI 2-sided [22.2 to 118.5]
Statistical Analysis 5: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 8 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 43.91, 95% CI 2-sided [21.0 to 66.8]
Statistical Analysis 6: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 8 - Adolescents; Test type: Other; p = 0.063, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 38.11, 95% CI 2-sided [-2.2 to 78.4]
Statistical Analysis 7: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 12 - Children; Test type: Other; p = 0.008, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 29.05, 95% CI 2-sided [8.2 to 49.9]
Statistical Analysis 8: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 12 - Adolescents; Test type: Other; p = 0.009, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 43.04, 95% CI 2-sided [11.9 to 74.2]
Statistical Analysis 9: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.006, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 44.20, 95% CI 2-sided [13.2 to 75.2]
Statistical Analysis 10: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.003, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 81.37, 95% CI 2-sided [30.4 to 132.3]
Statistical Analysis 11: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 36 - Children; Test type: Other; p = 0.004, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 58.49, 95% CI 2-sided [19.8 to 97.2]
Statistical Analysis 12: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 36 - Adolescents; Test type: Other; p = 0.039, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 50.90, 95% CI 2-sided [2.7 to 99.1]
Statistical Analysis 13: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 52 - Children; Test type: Other; p = 0.002, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 53.76, 95% CI 2-sided [21.7 to 85.8]
Statistical Analysis 14: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 52 - Adolescents; Test type: Other; p = 0.057, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 49.13, 95% CI 2-sided [-1.6 to 99.8]

12. Secondary Outcome: Change From Baseline in Average Morning Catheterized Volume
Description: The first morning catheterized volume was the first recorded non-zero volume within or after the hour of the wake-up time on a volume-measuring day in the e-diary. The average first morning catheterized volume was calculated as the average of the available first morning catheterized volumes recorded for the 2 measuring days in the weekend e-diary, whether or not these 2 days were consecutive. If the first morning catheterized volume was recorded on 1 single day of the weekend e-diary, the average morning catheterized is the first morning catheterized that day. If no first morning catheterized volumes are recorded on any day of the weekend e-diary, the average first morning catheterized volume was missing. A valid bladder diary day in the weekend diary was any e-diary day for which >=1 catheterized volume >0 mL was recorded with complete date and time.
Time Frame: Baseline and weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 41 | 21
mL
  Change at Week 2 | 7.98 (101.36) | 39.52 (80.24)
  Change at Week 4: number analyzed (Participants) | 40 | 20
  Change at Week 4 | 19.81 (89.04) | 75.25 (105.72)
  Change at Week 8 | 34.01 (89.53) | 44.43 (89.01)
  Change at Week 12: number analyzed (Participants) | 39 | 21
  Change at Week 12 | 8.68 (80.16) | 38.23 (66.80)
  Change at Week 24: number analyzed (Participants) | 36 | 20
  Change at Week 24 | 40.76 (116.41) | 86.66 (96.55)
  Change at Week 36: number analyzed (Participants) | 37 | 21
  Change at Week 36 | 31.08 (145.63) | 68.47 (122.43)
  Change at Week 52: number analyzed (Participants) | 39 | 21
  Change at Week 52 | 31.83 (94.25) | 38.14 (108.06)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 2 - Children; Test type: Other; p = 0.617, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 7.98, 95% CI 2-sided [-24.0 to 40.0]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 2 - Adolescents; Test type: Other; p = 0.035, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 39.52, 95% CI 2-sided [3.0 to 76.0]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p = 0.167, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 19.81, 95% CI 2-sided [-8.7 to 48.3]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.005, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 75.25, 95% CI 2-sided [25.8 to 124.7]
Statistical Analysis 5: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 8 - Children; Test type: Other; p = 0.020, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 34.01, 95% CI 2-sided [5.7 to 62.3]
Statistical Analysis 6: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 8 - Adolescents; Test type: Other; p = 0.033, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 44.43, 95% CI 2-sided [3.9 to 84.9]
Statistical Analysis 7: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 12 - Children; Test type: Other; p = 0.503, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 8.68, 95% CI 2-sided [-17.3 to 34.7]
Statistical Analysis 8: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 12 - Adolescents; Test type: Other; p = 0.016, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 38.23, 95% CI 2-sided [7.8 to 68.6]
Statistical Analysis 9: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.043, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 40.76, 95% CI 2-sided [1.4 to 80.2]
Statistical Analysis 10: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 86.66, 95% CI 2-sided [41.5 to 131.8]
Statistical Analysis 11: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 36 - Children; Test type: Other; p = 0.203, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 31.08, 95% CI 2-sided [-17.5 to 79.6]
Statistical Analysis 12: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 36 - Adolescents; Test type: Other; p = 0.019, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 68.47, 95% CI 2-sided [12.7 to 124.2]
Statistical Analysis 13: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 52 - Children; Test type: Other; p = 0.042, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 31.83, 95% CI 2-sided [1.3 to 62.4]
Statistical Analysis 14: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 52 - Adolescents; Test type: Other; p = 0.121, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 38.14, 95% CI 2-sided [-11.0 to 87.3]

13. Secondary Outcome: Change From Baseline in Mean Number of Leakage Episodes Per Day
Description: For each participant, the mean number of leakage episodes per day (during day & night time) was calculated using all available/non-missing number of leakage episodes for the 2 measuring days in the weekend diary during day & night time. If the number of leakage episodes was recorded on 1 single day in the 7-day diary during day & night time, the mean number of leakage episodes per day during day & night time is equal to the total number of leakage episodes recorded that day during day & night time. If no leakage episodes were recorded on any day of the weekend diary during day & night time, the mean number of leakage episodes per day was zero. Participants who did not report any leakage episode during the visit were imputed with a '0' for that visit. A valid bladder diary day in the weekend diary was any e-diary day for which ≥1 catheterized volume >0 mL was recorded with complete date and time.
Time Frame: Baseline and weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: leakage episodes per day
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 39 | 17
leakage episodes per day
  Change at Week 2 | 0.35 (9.35) | -0.53 (1.30)
  Change at Week 4: number analyzed (Participants) | 36 | 15
  Change at Week 4 | -1.14 (3.39) | -0.87 (1.68)
  Change at Week 8: number analyzed (Participants) | 35 | 10
  Change at Week 8 | 1.16 (16.11) | -0.65 (1.78)
  Change at Week 12: number analyzed (Participants) | 33 | 13
  Change at Week 12 | 0.37 (13.03) | -0.65 (1.55)
  Change at Week 24: number analyzed (Participants) | 31 | 14
  Change at Week 24 | 0.18 (10.05) | -0.75 (1.28)
  Change at Week 36: number analyzed (Participants) | 30 | 13
  Change at Week 36 | -1.98 (4.33) | -0.81 (1.47)
  Change at Week 52: number analyzed (Participants) | 32 | 13
  Change at Week 52 | -0.94 (2.96) | -1.12 (1.97)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 2 - Children; Test type: Other; p = 0.818, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.35, 95% CI 2-sided [-2.7 to 3.4]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 2 - Adolescents; Test type: Other; p = 0.114, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -0.53, 95% CI 2-sided [-1.2 to 0.1]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p = 0.052, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -1.14, 95% CI 2-sided [-2.3 to 0.0]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.066, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -0.87, 95% CI 2-sided [-1.8 to 0.1]
Statistical Analysis 5: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 8 - Children; Test type: Other; p = 0.674, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.16, 95% CI 2-sided [-4.4 to 6.7]
Statistical Analysis 6: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 8 - Adolescents; Test type: Other; p = 0.278, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -0.65, 95% CI 2-sided [-1.9 to 0.6]
Statistical Analysis 7: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 12 - Children; Test type: Other; p = 0.871, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.37, 95% CI 2-sided [-4.2 to 5.0]
Statistical Analysis 8: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 12 - Adolescents; Test type: Other; p = 0.153, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -0.65, 95% CI 2-sided [-1.6 to 0.3]
Statistical Analysis 9: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.922, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.18, 95% CI 2-sided [-3.5 to 3.9]
Statistical Analysis 10: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.047, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -0.75, 95% CI 2-sided [-1.5 to 0.0]
Statistical Analysis 11: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 36 - Children; Test type: Other; p = 0.018, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -1.98, 95% CI 2-sided [-3.6 to -0.4]
Statistical Analysis 12: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 36 - Adolescents; Test type: Other; p = 0.070, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -0.81, 95% CI 2-sided [-1.7 to 0.1]
Statistical Analysis 13: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 52 - Children; Test type: Other; p = 0.083, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -0.94, 95% CI 2-sided [-2.0 to 0.1]
Statistical Analysis 14: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 52 - Adolescents; Test type: Other; p = 0.064, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -1.12, 95% CI 2-sided [-2.3 to 0.1]

14. Secondary Outcome: Change From Baseline in Mean Number of Leakage Episodes Per Day: Updated Analysis
Description: For each participant, the mean number(no.) of leakage episodes per day (during day & night time) was calculated using all available/non-missing no. of leakage episodes for the 2 measuring days in the weekend diary during day & night time. If the no. of leakage episodes was recorded on 1 single day in the 7-day diary during day & night time, the mean no. of leakage episodes per day during day & night time is equal to the total no. of leakage episodes recorded that day during day & night time. If no leakage episodes were recorded on any day of the weekend diary during day & night time, the mean no. of leakage episodes per day was zero. Participants who did not report leakage episode during the visit were imputed with a '0' for that visit. A valid bladder diary day in weekend diary was any e-diary day for which ≥1 catheterized volume >0 mL was recorded with complete date and time. Updated analysis is presented because one participant entered weight of leakage instead of no. of leakages.
Time Frame: Baseline and weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: leakage episodes per day
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 30 | 21
leakage episodes per day
  Change at Week 2 | 0.78 (10.63) | -0.71 (1.27)
  Change at Week 4: number analyzed (Participants) | 29 | 21
  Change at Week 4 | -1.32 (3.63) | -0.95 (1.48)
  Change at Week 8: number analyzed (Participants) | 29 | 19
  Change at Week 8 | 1.68 (17.70) | -0.84 (1.40)
  Change at Week 12: number analyzed (Participants) | 28 | 21
  Change at Week 12 | 0.49 (14.23) | -0.86 (1.22)
  Change at Week 24: number analyzed (Participants) | 27 | 21
  Change at Week 24 | -2.34 (3.66) | -0.98 (1.08)
  Change at Week 36: number analyzed (Participants) | 26 | 21
  Change at Week 36 | -4.10 (9.92) | -0.98 (1.25)
  Change at Week 52: number analyzed (Participants) | 27 | 21
  Change at Week 52 | -1.99 (3.49) | -1.05 (1.61)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 2 - Children; Test type: Other; p = 0.692, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 2 - Adolescents; Test type: Other; p = 0.018, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p = 0.061, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.008, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 5: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 8 - Children; Test type: Other; p = 0.612, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 6: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 8 - Adolescents; Test type: Other; p = 0.018, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 7: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 12 - Children; Test type: Other; p = 0.858, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 8: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 12 - Adolescents; Test type: Other; p = 0.004, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 9: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.003, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 10: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 11: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 36 - Children; Test type: Other; p = 0.045, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 12: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 36 - Adolescents; Test type: Other; p = 0.002, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 13: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 52 - Children; Test type: Other; p = 0.006, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0
Statistical Analysis 14: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 52 - Adolescents; Test type: Other; p = 0.007, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0

15. Secondary Outcome: Change From Baseline in Number of Dry Days Per 7 Days (Day and Night Time)
Description: Dry days were defined as leakage-free days, this included day and night time. Participants recorded dry days in the 7-day diary. Dry days were calculated as follows: Ddry was the number of valid diary days where the response to the question 'Did you leak between this catheterization and the last one' was 'No' each time a new catheterization was entered in the e-diary during the day & night time period. Dwet was the number of valid diary days where the response to the question 'Did you leak between this catheterization and the last one' was 'Yes' for at least one catheterization entered during the day and night time period. If (Ddry + Dwet) > 3, the number of dry days per 7 days was calculated as Ddry/(Ddry + Dwet) x 7, otherwise the value was missing.
Time Frame: Baseline and weeks 2, 4, 8, 12, 24, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dry days per 7 days
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 43 | 24
dry days per 7 days
  Change at Week 2 | 0.34 (0.91) | 0.82 (1.90)
  Change at Week 4: number analyzed (Participants) | 42 | 24
  Change at Week 4 | 0.68 (1.69) | 1.36 (1.91)
  Change at Week 8: number analyzed (Participants) | 43 | 23
  Change at Week 8 | 1.14 (2.15) | 2.26 (2.48)
  Change at Week 12 | 1.31 (2.50) | 1.93 (2.46)
  Change at Week 24: number analyzed (Participants) | 41 | 24
  Change at Week 24 | 1.34 (2.18) | 2.17 (2.38)
  Change at Week 36: number analyzed (Participants) | 39 | 24
  Change at Week 36 | 1.33 (2.43) | 1.88 (2.13)
  Change at Week 52: number analyzed (Participants) | 40 | 24
  Change at Week 52 | 1.38 (2.65) | 2.14 (2.51)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 2 - Children; Test type: Other; p = 0.018, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.34, 95% CI 2-sided [0.1 to 0.6]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 2 - Adolescents; Test type: Other; p = 0.045, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.82, 95% CI 2-sided [0.0 to 1.6]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 4 - Children; Test type: Other; p = 0.013, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.68, 95% CI 2-sided [0.1 to 1.2]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 4 - Adolescents; Test type: Other; p = 0.002, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.36, 95% CI 2-sided [0.6 to 2.2]
Statistical Analysis 5: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 8 - Children; Test type: Other; p = 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.14, 95% CI 2-sided [0.5 to 1.8]
Statistical Analysis 6: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 8 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 2.26, 95% CI 2-sided [1.2 to 3.3]
Statistical Analysis 7: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 12 - Children; Test type: Other; p = 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.31, 95% CI 2-sided [0.5 to 2.1]
Statistical Analysis 8: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 12 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.93, 95% CI 2-sided [0.9 to 3.0]
Statistical Analysis 9: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.34, 95% CI 2-sided [0.7 to 2.0]
Statistical Analysis 10: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 2.17, 95% CI 2-sided [1.2 to 3.2]
Statistical Analysis 11: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 36 - Children; Test type: Other; p = 0.002, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.33, 95% CI 2-sided [0.5 to 2.1]
Statistical Analysis 12: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 36 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.88, 95% CI 2-sided [1.0 to 2.8]
Statistical Analysis 13: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 52 - Children; Test type: Other; p = 0.002, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.38, 95% CI 2-sided [0.5 to 2.2]
Statistical Analysis 14: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 52 - Adolescents; Test type: Other; p < 0.001, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 2.14, 95% CI 2-sided [1.1 to 3.2]

16. Secondary Outcome: Change From Baseline in Pediatric Incontinence Questionnaire (PIN-Q) Score
Description: PIN-Q measured quality of life via an e-diary. Total score ranged from 0 (no effect) to 80 (worst effect); decrease in score indicated improvement. Total score was 20x average of individual PinQ items, the 20 Likert scales were converted to a score: Items 6 & 17; 0: "No" to 4: "Definitely" was used; & For the other 18 items; 0: "No" to 4: "All the time" was used. Expectation that questionnaires had limited missing values; if answers >2 questions were missing, total score was not calculated & was missing. Individual item scores were directly imputed. Change from baseline to each post-baseline visit in the total score was post-baseline visit value minus baseline value. If either baseline or post-baseline visit value was missing, change from baseline was missing. If change was: <0, improvement between 2 time-points; =0, no change between 2 time points; >0, worsening between 2 time points.
Time Frame: Baseline and weeks 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 24 | 21
units on a scale
  Change at Week 24 | 2.04 (10.53) | -4.90 (14.13)
  Change at Week 52: number analyzed (Participants) | 23 | 19
  Change at Week 52 | 1.30 (12.17) | -6.79 (14.50)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.352, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 2.04, 95% CI 2-sided [-2.40 to 6.49]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.127, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -4.90, 95% CI 2-sided [-11.34 to 1.53]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 52 - Children; Test type: Other; p = 0.613, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 1.30, 95% CI 2-sided [-3.96 to 6.57]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 52 - Adolescents; Test type: Other; p = 0.056, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = -6.79, 95% CI 2-sided [-13.78 to 0.20]

17. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity Scale (PGI-S)
Description: The PGI-S was an answer to the question: "How did you feel about your bladder condition during the past 3 days?" Participants evaluated their recent condition as "Really Bad"(0), "Bad" (1), "Not Bad, Not Good" (2), "Good" (3) &"Really Good" (4). An increase indicated improvement. The total score ranged from 0 to 4, where higher scores indicated improvement.The change from baseline to each postbaseline visit in the PGI-S score is the value at the post-baseline visit minus the value at the baseline visit. If either the baseline or the post-baseline visit value is missing, the change from baseline was missing. A positive change indicated an improvement while a negative change indicated a worsening.
Time Frame: Baseline and weeks 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 25 | 22
units on a scale
  Change at Week 24 | 0.36 (1.22) | 0.64 (1.00)
  Change at Week 52: number analyzed (Participants) | 24 | 19
  Change at Week 52 | 0.42 (1.21) | 0.95 (1.18)
Statistical Analysis 1: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 24 - Children; Test type: Other; p = 0.153, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.36, 95% CI 2-sided [-0.14 to 0.86]
Statistical Analysis 2: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 24 - Adolescents; Test type: Other; p = 0.007, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.64, 95% CI 2-sided [0.19 to 1.08]
Statistical Analysis 3: Comparison: Children (3 to < 12 Years); Change From Baseline at Week 52 - Children; Test type: Other; p = 0.106, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.42, 95% CI 2-sided [-0.10 to 0.93]
Statistical Analysis 4: Comparison: Adolescents (12 to < 18 Years); Change From Baseline at Week 52 - Adolescents; Test type: Other; p = 0.003, t-test, 2 sided — From a 2-sided paired t-test, testing the null hypothesis that change from baseline is equal to 0; Mean Difference (Net) = 0.95, 95% CI 2-sided [0.38 to 1.51]

18. Secondary Outcome: Number of Participants With Clinician Global Impression of Change (CGI-C)
Description: The Clinician Global Impression of Change (CGI-C) is a 7 point scale that required the clinician to assess how much the participant's overall bladder symptoms since the start of the study on day 1 has improved or worsened and rated as: very much improved (1); much improved (2); minimally improved (3); no change (4); minimally worse (5); much worse (6); or very much worse (7). The total score range from 1-7, where lower scores indicated improvement.
Time Frame: Weeks 24 and 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 41 | 24
Participants
  Week 24 - Very much Improved | 6 | 10
  Week 24 - Much Improved | 24 | 7
  Week 24 - Minimally Improved | 6 | 5
  Week 24 - No Change | 4 | 1
  Week 24 - Minimally Worse | 1 | 1
  Week 24 - Much Worse | 0 | 0
  Week 24 - Very Much Worse | 0 | 0
  Week 52 - Very Much Improved: number analyzed (Participants) | 38 | 23
  Week 52 - Very Much Improved | 8 | 9
  Week 52 - Much Improved: number analyzed (Participants) | 38 | 23
  Week 52 - Much Improved | 23 | 12
  Week 52 - Minimally Improved: number analyzed (Participants) | 38 | 23
  Week 52 - Minimally Improved | 5 | 1
  Week 52 - No Change: number analyzed (Participants) | 38 | 23
  Week 52 - No Change | 2 | 0
  Week 52 - Minimally Worse: number analyzed (Participants) | 38 | 23
  Week 52 - Minimally Worse | 0 | 0
  Week 52 - Much Worse: number analyzed (Participants) | 38 | 23
  Week 52 - Much Worse | 0 | 1
  Week 52 - Very Much Worse: number analyzed (Participants) | 38 | 23
  Week 52 - Very Much Worse | 0 | 0

19. Secondary Outcome: Number of Participants With Study Drug Acceptability for Tablets at Week 4
Description: Participants evaluated the taste of the study medication/tablets by ticking 1 of the following categories: "Really Bad" (0), "Bad" (1), "Not Bad, Not Good" (2), "Good" (3) & "Really Good" (4). Participants evaluated the swallow of the study medication/tablets by ticking one of the following categories: "Really Difficult" (0), "Difficult" (1), "Not Difficult, Not Easy" (2), "Easy" (3) and "Really Easy" (4).
Time Frame: Week 4
Population: The analysis population consisted of the FAS. Here, Overall Number of participants analyzed signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 9 | 12
Participants
  Taste - Really bad | 0 | 0
  Taste - Bad | 0 | 0
  Taste - Not bad, not good | 5 | 7
  Taste - Good | 3 | 4
  Taste - Really good | 1 | 1
  Swallow - Really difficult | 0 | 0
  Swallow - Difficult | 0 | 0
  Swallow - Not difficult, not easy | 1 | 0
  Swallow - Easy | 3 | 7
  Swallow - Really easy | 5 | 5

20. Secondary Outcome: Number of Participants With Study Drug Acceptability for Tablets at Week 24
Description: as for outcome 19
Time Frame: Week 24
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 17 | 23
Participants
  Taste - Really bad | 1 | 0
  Taste - Bad | 2 | 0
  Taste - Not bad, not good | 6 | 15
  Taste - Good | 4 | 6
  Taste - Really good | 4 | 2
  Swallow - Really difficult | 0 | 0
  Swallow - Difficult | 0 | 0
  Swallow - Not difficult, not easy | 2 | 2
  Swallow - Easy | 3 | 10
  Swallow - Really easy | 12 | 11

21. Secondary Outcome: Number of Participants With Study Drug Acceptability for Tablets at Week 52
Description: as for outcome 19
Time Frame: Week 52
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 17 | 20
Participants
  Taste - Really bad | 0 | 0
  Taste - Bad | 0 | 0
  Taste - Not bad, not good | 8 | 16
  Taste - Good | 6 | 2
  Taste - Really good | 3 | 2
  Swallow - Really difficult | 0 | 0
  Swallow - Difficult | 0 | 0
  Swallow - Not difficult, not easy | 2 | 2
  Swallow - Easy | 4 | 7
  Swallow - Really easy | 11 | 11

22. Secondary Outcome: Number of Participants With Study Drug Acceptability for Oral Suspension at Week 4
Description: Participants evaluated the taste of the study medication/oral suspension by ticking 1 of the following categories:"Really Bad" (0), "Bad" (1), "Not Bad, Not Good" (2), "Good" (3) & "Really Good" (4). Participants evaluated the smell of the study medication/oral suspension by ticking 1 of the following categories: "Really Bad" (0), "Bad" (1),"Not Bad, Not Good" (2), "Good" (3) & "Really Good" (4). Participants evaluated the consumption and the preparation of the study medication/oral suspension by ticking 1 of the following categories: "Really Difficult" (0),"Difficult" (1), "Not Difficult, Not Easy" (2), "Easy" (3) & "Really Easy" (4).
Time Frame: Week 4
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 22 | 2
Participants
  Taste - Really bad | 1 | 0
  Taste - Bad | 3 | 0
  Taste - Not bad, not good | 4 | 2
  Taste - Good | 11 | 0
  Taste - Really good | 3 | 0
  Smell - Really bad | 0 | 0
  Smell - Bad | 1 | 0
  Smell - Not bad, not good | 8 | 1
  Smell - Good | 12 | 1
  Smell - Really good | 1 | 0
  Take - Really difficult | 0 | 0
  Take - Difficult | 0 | 0
  Take - Not difficult, not easy | 4 | 0
  Take - Easy | 7 | 1
  Take - Really Easy | 11 | 1
  Prepare - Really difficult | 0 | 0
  Prepare - Difficult | 0 | 0
  Prepare - Not difficult, not easy | 2 | 0
  Prepare - Easy | 12 | 0
  Prepare - Really Easy | 8 | 2

23. Secondary Outcome: Number of Participants With Study Drug Acceptability for Oral Suspension at Week 24
Description: as for outcome 22
Time Frame: Week 24
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 23 | 2
Participants
  Taste - Really bad | 3 | 0
  Taste - Bad | 1 | 0
  Taste - Not bad, not good | 3 | 2
  Taste - Good | 10 | 0
  Taste - Really good | 6 | 0
  Smell - Really bad | 2 | 0
  Smell - Bad | 0 | 0
  Smell - Not bad, not good | 8 | 2
  Smell - Good | 11 | 0
  Smell - Really good | 2 | 0
  Take - Really difficult | 0 | 0
  Take - Difficult | 2 | 0
  Take - Not difficult, not easy | 2 | 0
  Take - Easy | 6 | 0
  Take - Really Easy | 13 | 2
  Prepare - Really difficult | 0 | 0
  Prepare - Difficult | 1 | 0
  Prepare - Not difficult, not easy | 3 | 0
  Prepare - Easy | 10 | 2
  Prepare - Really Easy | 9 | 0

24. Secondary Outcome: Number of Participants With Study Drug Acceptability for Oral Suspension at Week 52
Description: as for outcome 22
Time Frame: Week 52
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 22 | 2
Participants
  Taste - Really bad | 1 | 0
  Taste - Bad | 2 | 0
  Taste - Not bad, not good | 5 | 2
  Taste - Good | 8 | 0
  Taste - Really good | 6 | 0
  Smell - Really bad | 2 | 0
  Smell - Bad | 1 | 0
  Smell - Not bad, not good | 5 | 1
  Smell - Good | 12 | 1
  Smell - Really good | 2 | 0
  Take - Really difficult | 0 | 0
  Take - Difficult | 1 | 0
  Take - Not difficult, not easy | 3 | 0
  Take - Easy | 7 | 0
  Take - Really Easy | 11 | 2
  Prepare - Really difficult | 0 | 0
  Prepare - Difficult | 0 | 0
  Prepare - Not difficult, not easy | 3 | 0
  Prepare - Easy | 9 | 2
  Prepare - Really Easy | 10 | 0

25. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who was given the study drug or who had undergone study procedures and did not necessarily have a causal relationship with this treatment. An AE could therefore be any unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A treatment-emergent adverse event (TEAE) was defined as any AE with date of onset occurring on or after the first dose of study medication and up to the end of study.
Time Frame: From the first dose of study drug administration up to end-of-treatment (EoT) (up to week 52)
Population: The analysis population consisted of the safety analysis set (SAF), which included of all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
Number analyzed (Participants) | 55 | 31
Participants
  TEAE | 33 | 18
  Drug-related TEAE | 8 | 6
  Serious TEAE | 9 | 5
  Drug-related Serious TEAE | 0 | 0
  TEAE Leading to Death | 0 | 0
  Drug-related TEAE Leading to Death | 0 | 0
  TEAE Leading to Permanent Discontinuation | 3 | 0
  Drug-related TEAE Leading to Permanent Disc. | 2 | 0
  Death | 0 | 0

26. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Mirabegron
Description: Cmax was defined as the maximum plasma concentration of mirabegron.
Time Frame: A total of 4 samples were collected over 2 sampling days at 2 separate visits at any of week 4, 8, 12, 24, 36, or 52, at the following time points: Sampling day 1- Predose; Sampling day 2- Predose and 2 samples 2-5 hours postdose more than 1 hour apart.
Population: The analysis population consisted of the pharmacokinetic analysis set (PKAS), which consisted of the subset of the SAF for whom plasma concentration data were available to facilitate derivation of ≥ 1 pharmacokinetic parameter and for whom the time of the last dose prior to sampling was known.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Groups:
- Children PED25 (PKAS): Participants aged 3 to < 12 years who received pediatric equivalent dose of 25 mg at the time of PK sampling.
- Adolescents PED25 (PKAS): Participants aged 12 to < 18 years who received pediatric equivalent dose of 25 mg at the time of PK sampling.
- Children PED50 (PKAS): Participants aged 3 to < 12 years who received pediatric equivalent dose of 50 mg at the time of PK sampling.
- Adolescents PED50 (PKAS): Participants aged 12 to < 18 years who received pediatric equivalent dose of 50 mg at the time of PK sampling.
Arm/Group | Children PED25 (PKAS) | Adolescents PED25 (PKAS) | Children PED50 (PKAS) | Adolescents PED50 (PKAS)
Number analyzed (Participants) | 1 | 3 | 43 | 24
nanogram/milliliter (ng/mL) | 9.386 (NA) — Due to low number of participants, standard deviation could not be calculated. | 9.044 (5.407) | 20.55 (13.63) | 18.40 (12.45)

27. Secondary Outcome: Time to Reach Maximum Plasma Concentration of Mirabegron Following Drug Administration (Tmax)
Description: Tmax was defined as the time to reach maximum plasma concentration following drug administration.
Time Frame: as for outcome 26
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Children PED25 (PKAS) | Adolescents PED25 (PKAS) | Children PED50 (PKAS) | Adolescents PED50 (PKAS)
Number analyzed (Participants) | 1 | 3 | 43 | 24
hours | 3.000 (NA) — Due to low number of participants, data could not be calculated. | 3.500 (0.433) | 3.419 (0.6608) | 3.635 (1.101)

28. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC24) for Mirabegron
Description: AUC (0-24) is the area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours post-dose.
Time Frame: as for outcome 26
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter
Arm/Group | Children PED25 (PKAS) | Adolescents PED25 (PKAS) | Children PED50 (PKAS) | Adolescents PED50 (PKAS)
Number analyzed (Participants) | 1 | 3 | 43 | 24
nanogram*hour/milliliter | 166.3 (NA) — Due to low number of participants, standard deviation could not be calculated. | 137.8 (53.07) | 310.1 (163.1) | 291.6 (171.8)

29. Secondary Outcome: Plasma Concentration of Mirabegron at the End of a Dosing Interval at Steady State (Ctrough)
Description: Ctrough was defined as the measured plasma concentration of mirabegron at the end of a dosing interval at steady state.
Time Frame: as for outcome 26
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Children PED25 (PKAS) | Adolescents PED25 (PKAS) | Children PED50 (PKAS) | Adolescents PED50 (PKAS)
Number analyzed (Participants) | 1 | 3 | 43 | 24
ng/mL | 5.312 (NA) — Due to low number of participants, standard deviation could not be calculated. | 4.114 (1.186) | 9.024 (5.149) | 8.888 (5.588)

30. Secondary Outcome: Apparent Total Clearance of Mirabegron From Plasma After Oral Administration (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: as for outcome 26
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: Liter/hour (L/hr)
Arm/Group | Children PED25 (PKAS) | Adolescents PED25 (PKAS) | Children PED50 (PKAS) | Adolescents PED50 (PKAS)
Number analyzed (Participants) | 1 | 3 | 43 | 24
Liter/hour (L/hr) | 192.5 (NA) — Due to low number of participants, standard deviation could not be calculated. | 202.3 (83.05) | 230.9 (162) | 279.6 (294.2)

31. Secondary Outcome: Apparent Volume of Distribution After Non-intravenous Administration (Vz/F) of Mirabegron
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 26
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Children PED25 (PKAS) | Adolescents PED25 (PKAS) | Children PED50 (PKAS) | Adolescents PED50 (PKAS)
Number analyzed (Participants) | 1 | 3 | 43 | 24
Liter | 14450 (NA) — Due to low number of participants, standard deviation could not be calculated. | 15380 (6524) | 12150 (5630) | 14770 (6792)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to end-of-treatment (EoT) (up to week 52).
Arm/Group | Children (3 to < 12 Years) | Adolescents (12 to < 18 Years)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/31
Serious Adverse Events (participants affected / at risk) | 9/55 | 5/31
Other Adverse Events (participants affected / at risk) | 17/55 | 9/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children (3 to < 12 Years) (N=55) | Adolescents (12 to < 18 Years) (N=31)
Talipes (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Urethral perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Talipes correction (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children (3 to < 12 Years) (N=55) | Adolescents (12 to < 18 Years) (N=31)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 3 (5) | 5 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 4 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (6)
Urinary tract infection (Infections and infestations) | 4 (5) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 4 (5) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study after Sponsor publication of multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT02751931/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02751931/SAP_001.pdf